CLINICAL TRIAL: NCT04149925
Title: Improving Hemostasis in Sleeve Gastrectomy With Alternative Stapler
Brief Title: Endostapler Hemostasis Study
Status: Completed | Type: Observational
Sponsor: Lexington Medical Inc. (Industry)
Collaborators: Surgical Specialists of Louisiana (Other)
Responsible Party: Sponsor
Other Study IDs: Endostapler01
Record Dates: First submitted 2019-10-31; First posted 2019-11-04 (Actual); Results first posted 2020-04-08 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Intraoperative Staple Line Bleeding as Measured by the Provided Bleeding Severity Scale

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- AEON Endostapler: Stapling performed by AEON Endostapler
  Interventions: Device: AEON Endostapler
- Echelon Flex Powered Stapler: Stapling performed by Echelon Flex Powered Stapler
  Interventions: Device: Echelon Flex Powered Stapler

INTERVENTIONS:
Device: AEON Endostapler — Surgery with AEON Endostapler
  Groups: AEON Endostapler
Device: Echelon Flex Powered Stapler — Surgery with Echelon Flex Powered Stapler
  Groups: Echelon Flex Powered Stapler

SUMMARY:
The goal of this prospective, multi-center, post-market study is to measure AEON™ Endostapler performance with the EASY/THICK MODE feature for laparoscopic bariatric surgery against the Echelon Flex™ Powered Stapler system from Ethicon. Stapler performance will be evaluated primarily by incidence and degree of staple line bleeding through a third-party blinded primary outcome evaluator. The study will include 60 total consecutive cases of individuals undergoing a planned laparoscopic sleeve gastrectomy (LSG). The LSG procedure will be performed according to institutional standard-of-care and all subjects will undergo standard preoperative evaluation as well as post-operative care. Relevant data will be collected using the Data Collection sheet which should be filled out following each procedure by a member of the surgical or nursing team.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing planned laparoscopic sleeve gastrectomy with signed surgery consent form
* Informed consent for study obtained and signed from each subject

Exclusion Criteria:

* Planned open surgical approach
* Prior bariatric operation (i.e. revisional bariatric surgery)
* Use of staple line reinforcement material (buttress)
* Patients taking anticoagulants
* Patients under the age of 18 on the date of the surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: See above
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2020-01-24 (Actual); Study Completion 2020-02-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Avala Hospital, Covington, Louisiana
  - Crescent City Surgical Centre, Metairie, Louisiana
  - Southern Surgical Hospital, Slidell, Louisiana

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AEON Endostapler | Echelon Flex Powered Stapler
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AEON Endostapler | Echelon Flex Powered Stapler | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (11) | 45 (11) | 46 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 25 | 43
  Male | 12 | 5 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m^2] | 44 (6) | 46 (7) | 45 (7)

OUTCOME MEASURES:

1. Primary Outcome: Staple Line Bleeding
Description: Intraoperative staple line bleeding as measured by the provided bleeding severity scale (1: No bleeding; 2: Minimal bleeding; 3: Moderate bleeding; 4: Excessive bleeding; 5: Profuse bleeding)
Time Frame: 10 seconds after last staple line
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AEON Endostapler | Echelon Flex Powered Stapler
Number analyzed (Participants) | 30 | 30
score on a scale | 2.08 (.98) | 2.57 (1.13)
Statistical Analysis 1: Comparison: AEON Endostapler vs Echelon Flex Powered Stapler; Test type: Superiority; p = 0.01, t-test, 2 sided — Significant when p<0.05

2. Secondary Outcome: Staple Line Leaking
Description: Incidence of postoperative leakage during one-month monitoring period following procedure
Time Frame: 1 month following procedure
Measure: Count of Participants; unit: Participants
Arm/Group | AEON Endostapler | Echelon Flex Powered Stapler
Number analyzed (Participants) | 30 | 30
Participants
  Yes | 0 | 0
  No | 30 | 30

3. Secondary Outcome: Adverse Events
Description: Incidence of reported device-related adverse events
Time Frame: 1 month following procedure
Measure: Count of Participants; unit: Participants
Arm/Group | AEON Endostapler | Echelon Flex Powered Stapler
Number analyzed (Participants) | 30 | 30
Participants
  Yes | 0 | 0
  No | 30 | 30

4. Secondary Outcome: Product Malfunction
Description: Incidence of product malfunction during procedure
Time Frame: During surgery
Measure: Count of Participants; unit: Participants
Arm/Group | AEON Endostapler | Echelon Flex Powered Stapler
Number analyzed (Participants) | 30 | 30
Participants
  Yes | 0 | 0
  No | 30 | 30

5. Secondary Outcome: Blood Transfusion
Description: Incidence of intraoperative or postoperative blood transfusion within 72 hours of surgery start time
Time Frame: Within 72 hours of surgery start
Measure: Count of Participants; unit: Participants
Arm/Group | AEON Endostapler | Echelon Flex Powered Stapler
Number analyzed (Participants) | 30 | 30
Participants
  Yes | 0 | 0
  No | 30 | 30

6. Secondary Outcome: Pain Level
Description: Postoperative pain level as measured by a standard pain severity scale of 0-10 where 0 means no pain and 10 means severe pain.
Time Frame: 1 week following procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AEON Endostapler | Echelon Flex Powered Stapler
Number analyzed (Participants) | 30 | 30
score on a scale | 1.8 (2.9) | 1.6 (2.7)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | AEON Endostapler | Echelon Flex Powered Stapler
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2019-09-12): https://cdn.clinicaltrials.gov/large-docs/25/NCT04149925/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-09-09): https://cdn.clinicaltrials.gov/large-docs/25/NCT04149925/Prot_SAP_001.pdf